CLINICAL TRIAL: NCT01173224
Title: A Phase I C Clinical Study With Influenza Antiviral DAS181-F03: Double-Blind, Randomized, Placebo-Controlled, Single Dose and Multiple Dose Escalation Study in Healthy Adults
Brief Title: Influenza Antiviral DAS181-F03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-0104; N01AI80026C
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2012-11

CONDITIONS: Influenza
Keywords: influenza, DAS181, antiviral
MeSH Terms: conditions — Influenza, Human | interventions — oplunofusp

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Cohort 2: 20 mg 10 days (Experimental): Cohort 2: 20mg DAS181 or placebo for 10 consecutive days (total dose of 200mg).
  Interventions: Drug: Placebo; Drug: DAS181
- Cohort 3: 30 mg 1 day (Experimental): Cohort 3: 30mg DAS181 or placebo for 1 day (total dose of 30mg).
  Interventions: Drug: Placebo; Drug: DAS181
- Cohort 1: 20 mg, 1 day (Experimental): Cohort 1: 20mg DAS181 or placebo for 1 day (total dose of 20mg).
  Interventions: Drug: Placebo; Drug: DAS181

INTERVENTIONS:
Drug: Placebo — Placebo: Cohort 1: 20mg DAS181 or placebo for 1 day (total dose of 20mg). Cohort 2: 20mg DAS181 or placebo for 10 consecutive days (total dose of 200mg). Cohort 3: 30mg DAS181 or placebo for 1 day (total dose of 30mg).
Drug: DAS181 — DAS181 F03: Cohort 1: 20mg DAS181 or placebo for 1 day (total dose of 20mg). Cohort 2: 20mg DAS181 or placebo for 10 consecutive days (total dose of 200mg). Cohort 3: 30mg DAS181 or placebo for 1 day (total dose of 30mg).

SUMMARY:
Influenza (flu) is a common respiratory infection and often causes severe illness. Few drugs are currently approved to treat influenza. This research will test the safety of an experimental anti-influenza drug called DAS181 that is given through an inhaler. The purpose of this study is to evaluate the safety of this new medication and how the body reacts to it. Any side effects will be measured by symptoms, physical examination or laboratory studies. About 27 healthy men and women age 18-45, who meet screening requirements, will participate. Three separate groups will be enrolled, with approximately 9 subjects in each group. Cohort 1:20 mg DAS181 or placebo for 1 day (total dose of 20 mg). Cohort 2: 20 mg DAS181 or placebo for 10 consecutive days (total dose of 200 mg). Cohort 3: 30 mg DAS 181 or placebo for 1 day (total dose of 30 mg.) Procedures include blood samples, electrocardiograms (measures heart activity) and breathing tests.

DETAILED DESCRIPTION:
Influenza is typically caused by infection of two types of viruses, influenza virus A and influenza virus B. The host cell receptors for influenza A and B viruses are cell surface sialic acids (SA). The Actinomyces viscosus sialidase Catalytic Domain (AvCD) sialidase domain in DAS181 selectively cleaves sialic acids from the host cells, thereby rendering them inaccessible to the influenza viral particles that require sialic acids as receptors. By binding to the negatively charged glycosaminoglycans on the surface of airway epithelial cells, the cationic C-terminal Amphiregulin (AR) tag anchors DAS181 on the respiratory epithelium, thereby improving treatment potency and retention of the investigational drug on the airway surface. DAS181 is the first candidate in a new class of influenza therapeutics, viral receptor inactivator. The primary objective is to determine the safety and tolerability of DAS181 encapsulated dry powder compared to placebo when administered by oral inhalation using a dry powder inhaler (DPI) in healthy adults. The secondary objective of this study is to investigate the pharmacokinetic and immunologic profile of DAS181 encapsulated dry powder dose to dose and compared to placebo when administered by oral inhalation using a DPI in healthy adults. A total of 27 normal healthy male and female subjects (9 per cohort) 18 to 45 years of age at the time of screening will be included in this study. This study will be a double-blind, randomized, placebo-controlled study of a three cohorts. Cohort 1:20 mg DAS181 or placebo for 1 day (total dose of 20 mg). Cohort 2: 20 mg DAS181 or placebo for 10 consecutive days (total dose of 200 mg). Cohort 3: 30 mg DAS 181 or placebo for 1 day (total dose of 30 mg.) The study will proceed to the next stage of multiple daily doses based on meeting study defined criteria. Within each dose cohort of nine, subjects will be randomly assigned to DAS181 or placebo at 2:1 ratios. Subjects will be admitted to the inpatient clinic on the day prior to first dose (Day -1). The subjects in single dose cohorts (Cohort 1 and 3) will stay in the inpatient unit for dosing (Day 0) and one day after dosing (Day 1). Subjects in Cohort 1 will come back for follow-up visits on Study Days 2, 3, 7, 14, and 30 . Subjects in Cohort 3 will return on Days 2, 3, 4, 5, 8. 10, 16, and 30. The subjects in the 10-day, multiple-dose cohort (Cohort 2) will stay in the inpatient clinic from Day -1 to 1 and will be required to come back for follow-up visits on Days 2 - 7. They will be seen (and optionally readmitted) Days 8 - 10 and will be seen as outpatients Days 11, 13, 15, 17, 20, 22, 24, and 27. All subjects will be asked to return for an additional blood draw to conduct an immunogenicity test at 90 days post final dosing. Subjects will be trained in proper inhalation techniques prior to dosing using a low range inspiratory flow measurement device.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects in good health in the opinion of the site Principal Investigator (PI) or subinvestigator as determined by vital signs, medical history, and a physical exam.
* Subjects must be able to verbalize understanding of the consent form, provide written informed consent and verbalize willingness to complete study procedures.
* Be 18 to 45 years of age (inclusive), at the time of screening.
* Subjects must have a Body Mass Index (BMI) of 18.5-35.
* No recent history of smoking in the past six months regardless of clinical relevance.
* Electrocardiogram (ECG) with no clinically significant abnormalities recorded at screening visit: PR interval within 120 and 200 ms, QRS interval < 120 ms, and QTc interval less than or equal to 440 ms.
* Blood pressure within normal limits (systolic 90-140 mm Hg; diastolic 50-90 mm Hg) and heart rate between 45 and 100 beats per minute.
* Chest X-ray shows no clinically significant abnormalities.
* Peak Expiratory Flow Rate (PEFR) will be greater than 80 percent predicted and Forced Expiratory Volume in One Second (FEV1) will be greater than 80 percent predicted. Note: Only one baseline value for PEFR and FEV1 can be used to support inclusion criterion.
* Negative Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBSAg), and Hepatitis C Virus (HCV) antibody screening tests.
* Negative screening tests for: marijuana, cocaine metabolite, amphetamines, opiates, Phencyclidine (PCP), barbiturates, benzodiazepines and ethanol.
* Subjects with the following laboratory criteria within provided range:

  1. Hemoglobin
  2. White blood cell (WBC) and platelet count
  3. Alkaline Phosphatase (ALKP), total bilirubin, Alanine Aminotransferase (ALT),
  4. Serum glucose. Note: If a non-fasting glucose is performed and is abnormal, a fasting glucose measurement may be measured in its place. If this is within the provided range, then subject may be enrolled.
  5. Serum creatinine
  6. Activated partial thromboplastin time (APTT) and Fibrinogen
* Urine glucose and blood tested by dipstick urinalysis are negative. Urine protein tested by dipstick is negative or trace. Menstruating females failing inclusion due to positive urine dipstick blood may be retested following cessation of menses.
* Female subjects must be post-menopausal (one year or greater without menses), surgically incapable of childbearing, or agreeable to practicing abstinence or two effective methods of birth control during the study period and for 12 weeks after study product administration. Acceptable methods may include:

  1. intrauterine device
  2. spermicide
  3. barrier contraception
  4. hormonal contraception.
* A female subject must have had a negative serum pregnancy test during the screening visit and a negative urine pregnancy test within 24 hours of drug dosing.
* If male, agrees to use medically accepted form of contraception from time of enrollment to 12 weeks after study product administration.
* Agrees not to drink any products containing caffeine (e.g., coffee, tea, soda) for 24 hours before the inpatient visit and during the entire inpatient admission.
* Agrees not to drink alcohol or participate in strenuous physical activity or exercise from 24 hours prior to the inpatient admission through the Day 7 (Cohorts 1 and 3) or Day 17 (Cohort 2) follow-up visit.

Exclusion Criteria:

* Have received any investigational drug or vaccine within 30 days prior to study drug dosing or have had a serious adverse reaction or hypersensitivity to any drug.
* Is planning to participate in another clinical trial within 30 days after the last dose of DAS181. Have received blood products within 6 months of study enrollment.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Have been on a liquid protein diet in the last month.
* Are allergic or intolerant to lactose.
* Have sickle cell disease.
* Have used any prescription drugs, excluding hormonal contraception, within 7 days prior to admission. Non-prescription drugs or OTC drugs (including herbal supplements) are allowed unless they require intranasal or inhalation administration.
* Existence of any surgical, medical or laboratory condition that, in the judgment of the site PI or subinvestigator, might interfere with the safety, distribution, metabolism or excretion of the drug.
* Subjects with concurrent respiratory diseases (e.g., asthma, allergic rhinitis, chronic obstructive pulmonary disease, cystic fibrosis, emphysema, or anaphylaxis), requiring acute or chronic medication, as determined by the investigator through medical history evaluation and physical examination.
* Subjects who have experienced a previous episode of acute upper respiratory tract infection, pneumonia, otitis, bronchitis, or sinusitis within 2 weeks prior to screening.
* Subjects with concurrent sustained respiratory symptoms (runny nose, sore throat, sneezing, coughing, or wheezing).
* Subjects who have an oral temperature above 37.8 degrees Celsius (100 degrees Fahrenheit).
* Subjects with cancer or history of hematologic malignancy. Cancer is defined as any active neoplastic diseases excluding noninvasive basal cell carcinoma.
* Subjects who have a planned hospital admission for any cause and/or a planned surgical procedure within 30 days of initiation of the study.
* Female subjects who are pregnant or breast-feeding.
* Subjects who have donated or lost more than 500 mL of blood in the three months prior to screening or who plan to donate blood during study participation.
* Subjects who have clinically significant medical or psychological conditions that would compromise the subject's safety, influence the results of the study, affect the subject's ability to participate in the study, or impair the subject's ability to provide informed consent.
* Subjects who have a history of drug dependence, or psychiatric illness within 2 years of study enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple dose DAS181 treatment: adverse events, hematology, clinical chemistry, blood coagulation, haptoglobin, urinalysis, throat swab for bacterial culture, ECG, chest X-ray, and spirometric lung function. | Up to Day 90

SECONDARY OUTCOMES:
Blood samples to determine the pharmacokinetic profile of DAS 181. | Day 0 through Day 30.
Blood samples to determine the immunogenic profile of DAS 181. | Day 0 through Day 90.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland, United States